CLINICAL TRIAL: NCT05867303
Title: A Phase 1, First-in-Human, Multicenter, Open-Label Study to Evaluate the Safety, Tolerability, Pharmacokinetic, Immunogenetic and Efficacy of RC198 in Subjects With Locally Advanced Unresectable or Metastatic Solid Tumors
Brief Title: A RC198 Study in Subjects With Locally Advanced Unresectable or Metastatic Solid Tumors
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: RemeGen Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RC198-G001
Record Dates: First submitted 2023-04-17; First posted 2023-05-19 (Actual); Last update posted 2024-08-16 (Actual); Status verified 2024-08

CONDITIONS: Melanoma; Urothelial Carcinoma; Renal Cell Carcinoma; Non-small Cell Lung Cancer; Head and Neck Squamous Cell Carcinoma; Colorectal Carcinoma
Keywords: Locally advanced unresectable or metastatic solid tumors
MeSH Terms: conditions — Melanoma; Carcinoma, Transitional Cell; Carcinoma, Renal Cell; Carcinoma, Non-Small-Cell Lung; Squamous Cell Carcinoma of Head and Neck; Colorectal Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- RC198 Injection (Experimental): RC198 injection will be administered subcutaneously on Day 1 of Week 1 to Week 4 (inclusive) of each 6-week (42-day) cycle.
  Interventions: Drug: RC198 Injection

INTERVENTIONS:
Drug: RC198 Injection — RC198 injection will be administered subcutaneously on Day 1 of Week 1 to Week 4 (inclusive) of each 6-week (42-day) cycle.

SUMMARY:
Safety study of RC198 in Subjects with Solid Tumors.

DETAILED DESCRIPTION:
This is a Phase 1, first-in-human, open-label study to determine the safety, tolerability, maximum tolerated dose (MTD) and/or recommended Phase 2 dose (RP2D) of RC198 in subjects with locally advanced unresectable or metastatic solid tumors for whom standard therapy does not exist, is no longer effective, or is not acceptable.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects with the ability to understand and give written informed consent for participation in this trial, including all evaluations and procedures as specified by this protocol.
2. Subjects with locally advanced unresectable or metastatic solid tumors who experience disease progression after standard treatment, or unable to tolerate standard treatment, or refuse standard treatment.
3. At least 1 measurable or evaluable lesion per Response Evaluation Criteria In Solid Tumors (RECIST) v1.1.
4. Male or female aged ≥ 18 years.
5. ECOG PS score of 0 or 1.
6. Anticipated life expectancy of > 12 weeks.
7. Adequate bone marrow, liver, and renal function defined as:

   * Absolute neutrophil count ≥ 1.5× 109/L.
   * Absolute lymphocyte count ≥ 500/μL.
   * Platelet ≥ 100 × 109/L.
   * Hemoglobin ≥ 90 g/L without receiving erythropoietin (EPO), granulocyte colony stimulating factor (G-CSF), or granulocyte-macrophage colony stimulating factor (GM-CSF) within 14 days and blood transfusion including red blood cell and platelet transfusion in at least 7 days prior to first dose of investigational product.
   * Total bilirubin ≤ 1.5 × ULN or up to 3 × ULN if Gilbert syndrome.
   * Alanine aminotransaminase (ALT), aspartate aminotransferase (AST) ≤ 2.5 × ULN when there is no liver metastasis. ALT, AST ≤ 5 × ULN when there is liver metastasis
   * Serum creatinine ≤ 1.5 × ULN, or creatinine clearance ≥ 60 mL/min (using Cockcroft-Gault formula); Urine protein < 2 + or 24 hour total urine protein quantity < 1g.
   * Activated partial thromboplastin time (APTT) ≤ 1.5× ULN; international normalized ratio (INR) ≤ 1.5.
8. Left ventricular ejection fraction ≥ 50%, as determined by echocardiogram or multiple-gated acquisition (MUGA) scan.
9. Willingness to avoid pregnancy or fathering children based on the criteria below:

   1. Women of childbearing potential (WOCBP) who engage in heterosexual intercourse or male subjects whose sexual partners are WOCBP must be able to and agree to use an acceptable, highly effective, double barrier contraception commencing from Screening, during study, and for 6 months after the last dose of investigational product, including:

      * Simultaneous use of hormonal contraceptives and must agree to use the same hormonal contraceptive throughout the study, and a condom for the male partner.
      * Simultaneous use of intrauterine device (IUD) and condom for the male partner.
      * Simultaneous use of diaphragm or cervical cap and condom for the male partner.
      * Sterile male partner (vasectomized for at least 6 months prior to first dose of investigational product).
      * True abstinence, defined as no sexual intercourse (heterosexual couples). Periodic abstinence and withdrawal are not acceptable methods.

      Subjects with same-sex partners (abstinence from penile-vaginal intercourse) or who are abstinent from heterosexual intercourse are not required use contraception when this is their preferred and usual lifestyle.
   2. WOCBP must have a negative serum beta human-chorionic gonadotropin (β-hCG) pregnancy test at Screening and a negative pregnancy test on Day 1 of each cycle. In the event of a positive urine pregnancy test, a serum pregnancy test will be performed for confirmation.
   3. Must agree not to donate ova or sperm from Screening, during study, and for 6 months after the last dose of investigational product
   4. Must agree not to donate ova or sperm from Screening, during study, and for 6 months after the last dose of investigational product

Exclusion Criteria:

1. Pregnant or lactating.
2. Known to be human immunodeficiency virus (HIV) positive, with active hepatitis (HBV) characterized by elevated levels of HBV ribonucleic acid exceeding the ULN; or active hepatitis C (HCV) with positive HCV ribonucleic acid (RNA); Subjects who are Hepatitis B surface antigen positive or hepatitis B core antibody positive must have undetectable quantitative DNA polymerase chain reaction (PCR).
3. Administration of a live vaccine within 28 days before first dose of investigational and during the study. Note: Seasonal vaccines for influenza or Coronavirus Disease 2019 (COVID-19) vaccines are generally inactivated vaccines and are allowed. Intranasal vaccines are live vaccines and are not allowed.
4. Previous anti-tumor therapies (including surgery, chemotherapy, traditional Chinese medicine, radiotherapy, immunotherapy, biological therapy, hormonal therapy, or investigational agents for cancer treatment) within 4 weeks or within 5 half-lives of anti-tumor agents, whichever is shorter, prior to the first dose of investigational product, or palliative radiotherapy for bone metastases within 2 weeks prior to the first dose of investigational product.
5. Previous adverse reactions resulting from previous anti-tumor therapies, which have not resolved to Grade 0 or 1 according to NCI CTCAE v5.0 (except for alopecia, fatigue, pigmentation and other conditions with no safety risk according to Investigator's opinion) or Baseline within 4 weeks prior to first administration of the investigational product.
6. Experienced prior Grade 3 or higher immune-related toxicity that resulted in permanent drug discontinuation (subjects with prior temporary drug interruptions due to endocrinopathies etc. are eligible).
7. History of therapy with an agent targeting of IL-15 or IL-2.
8. Known hypersensitivity to any excipient contained in the drug formulation of investigational products or supplements to be administered during the study.
9. Uncontrolled diseases including:

   1. Uncontrolled infection requiring systematic antibiotics, antivirals or antifungals within 4 weeks prior to first administration of the investigational product.
   2. Active infection with COVID-19.
   3. Active tuberculosis infection, or still on anti-tuberculosis therapy or received anti-tuberculosis therapy within 1 year prior to first administration of the investigational product.
   4. Symptomatic congestive heart failure Grade II-IV (New York Heart Association [NYHA]), symptomatic or uncontrolled arrhythmias, QTc interval > 480 ms or personal or family history of congenital long/short QT syndrome, Severe or unstable angina pectoris, coronary or peripheral artery bypass grafting.
   5. Uncontrollable hypertension (systolic blood pressure ≥ 160mmHg or diastolic blood pressure ≥ 100mmHg).
   6. Systemic diseases, including diabetes pulmonary fibrosis, acute lung disease, interstitial lung disease, cirrhosis, etc.
10. History of any arterial thromboembolic event within 6 months prior to the first administration of investigational product, including myocardial infarction, unstable angina pectoris, pulmonary embolism, cerebrovascular stroke, or transient ischemic attack, etc.
11. History of deep vein thrombosis or any other severe thromboembolism within 3 months prior to the first administration of investigational product (implantable venous access port or catheter-derived thrombosis, or superficial venous thrombosis is not considered as "severe" thromboembolism).
12. History of life-threatening bleeding, or Grade 3 or 4 gastrointestinal/variceal bleeding requiring blood transfusion, endoscopy, or surgery, within 3 months prior to the first administration of investigational product.
13. History of other acquired/congenital immunodeficiency diseases.
14. History of organ transplantation allogeneic bone marrow transplantation, or autologous hematopoietic stem cell transplantation.
15. A condition requiring systemic treatment with either corticosteroids (> 10 mg daily prednisone equivalent) within 7 days or other immunosuppressive medication(s) within 14 days of the first dose of investigational product. Subjects using physiologic replacement doses of prednisone at ≤ 10 mg/day, or its equivalent, are eligible.
16. Active autoimmune diseases or history of autoimmune diseases that may relapse.

    Note: Subjects with the following diseases are not excluded:
    1. Controlled Type I diabetes.
    2. Hypothyroidism (provided it is managed with hormone replacement therapy only).
    3. Controlled celiac disease.
    4. Skin diseases not requiring systemic treatment (eg, vitiligo, psoriasis, alopecia).
    5. Any other disease that is not expected to recur in the absence of external triggering factors.
17. History or presence of metastatic brain tumors. Subjects with confirmed brain metastases are eligible for the study provided that they are asymptomatic and radiologically stable without the need for corticosteroid treatment >10 mg or seizure prophylaxis for ≥ 4 weeks prior to first dose of investigational product.
18. Have undergone major surgeries within 4 weeks prior to first dose of investigational product.
19. Uncontrollable pleural effusion, pericardial effusion, or ascites requiring frequent drainage within 7 days prior to first dose of investigational product.
20. Under the treatment of heparin (eg, low molecular weight heparin [LMWH]) or other anticoagulants such as warfarin when administered at a therapeutic dose. Participants using prophylactic doses of heparin (LMWH) are eligible.
21. Diagnosis of any other malignancy within 2 years prior to enrollment, except for the following if adequately treated:

    * Local basal cell or squamous cell carcinoma of the skin or related localized.
    * Non-melanoma skin cancer.
    * Carcinoma in situ of the breast or of the cervix.
    * Non-muscle invasive bladder cancer.
    * Low grade (Gleason 6 or below) prostate cancer undergoing surveillance with no plans for treatment intervention or previously fully resected.
22. History or presence of uncontrolled mental illness or drug abuse disorder in opinion of the Investigator.
23. The subject is expected to be non-compliant with critical study procedures and is not willing or able to adhere to the study requirements.
24. Subject is deemed inappropriate for this clinical study, or participation in this clinical study is deemed not in the best interest of the subject, at the discretion of the Investigator.
25. Other acute or chronic diseases or abnormal laboratory test that may: increase risk of study participation or investigational product administration, interfere with the interpretation of study results, and disqualify the subject for study participation in the Investigator's judgment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2023-06-05 (Actual); Primary Completion 2024-09-30 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
MTD based on number of dose-limiting toxicities (DLTs) | First 4 weeks (28 days) after first dose of study drug
  The maximum tolerated dose (MTD) will be assessed based on the number of patients experiencing DLTs, graded according to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) v5.0.
Determine Recommended Phase 2 Dose (RP2D) | Informed consent through 28 days after the last dose of study drug
  The RP2D may be selected based on the MTD following consultation with the safety monitoring committee with all available data.
Incidence of Adverse Events [Safety and tolerability] | Informed consent through 28 days after the last dose of study drug
  The adverse events occurring or worsening on or after the first dose of the study drug will be recorded.

SECONDARY OUTCOMES:
Time to maximum serum concentration [Tmax] | Day 1- Day 5 of Week 1 and Week 4, Day 1 of Week 2, Week 3, Week 5 and Week 6 during cycle 1, and Day 1 of Week 1 and Week 4 during subsequent cycles, and EOT (7 days within subject discontinued study drug)
  Tmax of RC198
Area under the serum concentration verus time curve [AUC] | Day 1- Day 5 of Week 1 and Week 4, Day 1 of Week 2, Week 3, Week 5 and Week 6 during cycle 1, and Day 1 of Week 1 and Week 4 during subsequent cycles, and EOT (7 days within subject discontinued study drug)
  AUC of RC198
Maximum serum Concentration [Cmax] | Day 1- Day 5 of Week 1 and Week 4, Day 1 of Week 2, Week 3, Week 5 and Week 6 during cycle 1, and Day 1 of Week 1 and Week 4 during subsequent cycles, and EOT (7 days within subject discontinued study drug)
  Cmax of RC198
Immunogenicity of RC198 | D1 of W1 and W3 during cycle 1, and D1 of W1 during subsequent cycles, and EOT (7 days within subject discontinued study drug)
  Incidence of anti-drug antibody (ADA) against RC198
Object Response Rate (ORR) | Screening, then every 6 weeks (±7 days) after Day 1 of Cycle 1 Week 1 until 14 days after the last dose of the study drug. Assessed up to 24 months.
  ORR will be determined according to Response Evaluation Criteria in Solid Tumours (RECIST) v1.1. The ORR is defined as the number of patients are either complete response (CR) or partial response (PR), relative to the number of patients belonging to the study of interest
Disease Control Rate (DCR) | Screening, then every 6 weeks (±7 days) after Day 1 of Cycle 1 Week 1 until 14 days after the last dose of the study drug. Assessed up to 24 months.
  DCR is the proportion of patients with disease control.
Duration of response (DoR) | From first partial response (PR) or complete response (CR) until disease progression or death, whichever occurs first. Assessed up to 24 months.
  DoR is defined, for patients with response, as the time from first documentation of response (CR or PR) to the date of first documentation of progression of disease or death due to any causes whichever occurs first.
Progression Free Survival (PFS) | From the first dose until documented disease progression or death, whichever occurs first. Assessed up to 24 months.
  PFS is defined as the time from the date of first administration to the date of the first documentation of progressive disease or death due to any cause, whichever occurs first.

CONTACTS AND LOCATIONS:
Locations (5):
- Australia (3):
  - ICON Cancer Centre Wesley, Auchenflower, Queensland
  - Southern Oncology Clinical Research Unit, Bedford Park, South Australia
  - Cabrini Hospital Malvern, Malvern, Victoria
- China (2):
  - Sun Yat-sen University Cancer Center, Guangzhou, Guangdong
  - Zhongnan Hospital of Wuhan University, Wuhan, Hubei